CLINICAL TRIAL: NCT03546153
Title: Phenotyping Chronic Low Back Pain Patients With Central Sensitization
Brief Title: Examining Effects of Aerobic Exercise on Pain Sensation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00141062
Record Dates: First submitted 2018-05-22; First posted 2018-06-06 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aerobic exercise program (Experimental): Participants will complete 12 week exercise program.
  Interventions: Behavioral: Aerobic exercise program

INTERVENTIONS:
Behavioral: Aerobic exercise program — Exercise program consists of training for 60 minutes, three times per week for 12 weeks. Participants will use a treadmill, Nu stepper/bike or elliptical to exercise.

SUMMARY:
By doing this study, researchers hope to learn effects of aerobic exercise on over activated nervous system in people with chronic low back pain.

DETAILED DESCRIPTION:
Chronic low back pain is a common condition in the world. About 85% of people with low back pain do not know the cause of their pain. This leads to ineffective treatments.

Recently, the idea of an over activated nervous system is thought to be one of the main reasons for chronic pain. Over activated nervous system means pain processing areas in the spine or brain might be more sensitive. Aerobic exercise, such as walking and cycling, is often used to decrease chronic pain. Aerobic exercise is a form of physical exercise that strengthen the heart and lungs in order to improve the body's utilization of oxygen.

The researchers want to examine if aerobic exercise is effective in decreasing over activation of the nervous system. Gaining a better understanding of effects of aerobic exercise on the nervous system may lead to more effective treatments for low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Lower back pain (LBP) for more than 3 months
* A minimal pain level of 3 on the 0-10 pain numerical rating scale (NRS) in the last 7 days
* Can read and understand English.

Exclusion Criteria:

* Nerve root compression that resulted in numbness or decrease in sensation in the areas for the pain sensitivity tests as reported by the subject
* cervical or thoracic pain as a main complaint
* spinal pathologies such as fracture, tumor, infection, and severe inflammation
* severe spinal deformity
* severe cardiovascular and neurological diseases
* cancer
* history of spinal surgery
* currently seeking active treatments for LBP other than medications
* resting blood pressure more than 160/90 mmHg 49
* currently taking blood thinning medications
* uncontrolled diabetes
* cannot have blood pressure taken
* participated in a similar trial in the past

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Pain sensitivity (Pressure pain threshold) | Change from Baseline (pre-treatment) to after completion of 3 months of aerobic exercise training (post-treatment)
  Sensitivity will be measured using a pressure algometer.
2011 FM survey | Change from Baseline (pre-treatment) to after completion of 3 months of aerobic exercise training (post-treatment)
  Sensitivity will be measured using the 2011 Fibromyalgia (FM) Survey Criteria. The survey includes widespread pain index and symptom severity scale. The total score is 31 and scores more than 13 is considered fibromyalgia positive, suggesting presence of central sensitization.
Opioid consumption | Change from Baseline (pre-treatment) to after completion of 3 months of aerobic exercise training (post-treatment)
  Use of opioids (dose, frequency, and duration) will be obtained by interviewing the subjects
Oswestry Disability Index | Change from Baseline (pre-treatment) to after completion of 3 months of aerobic exercise training (post-treatment)
  This questionnaire consists of questions related to daily functions and degrees to which back pain interferes with these functions. Each items is measured on a 6-point scale with a total possible score of 50. Higher numbers indicate greater disability.

SECONDARY OUTCOMES:
Pain Sensitivity (CPM test) | Change from Baseline (pre-treatment) to after completion of 3 months of aerobic exercise training (post-treatment)
  Measure of the functionality of descending inhibitory pain pathways with use of pressure algometry.
Fear Avoidance Belief Questionnaire | Change from Baseline (pre-treatment) to after completion of 3 months of aerobic exercise training (post-treatment)
  The survey has items related to fear about physical and work activities. Each item is scored from 0-6 points, with higher number indicating increased fear of activity or work.
Pain Catastrophizing Scale | Change from Baseline (pre-treatment) to after completion of 3 months of aerobic exercise training (post-treatment)
  PCS is a validated 13--item scale with questions related to catastrophizing behavior. Total score is 52 with higher scores indicating greater catastrophic thoughts.
Beck Depression Inventory | Change from Baseline (pre-treatment) to after completion of 3 months of aerobic exercise training (post-treatment)
  Beck depression questionnaire contains 21 multiple-choice depression related questions on a scale value of 0 to 3. Higher scores indicate greater depressive symptoms.
Beck Anxiety Inventory | Change from Baseline (pre-treatment) to after completion of 3 months of aerobic exercise training (post-treatment)
  Beck anxiety questionnaire contains 21 multiple-choice questions, each score 0 (not al all) to 3 (severely). Higher scores indicate greater anxiety symptoms.
Pittsburgh Sleep Quality Index | Change from Baseline (pre-treatment) to after completion of 3 months of aerobic exercise training (post-treatment)
  Pittsburgh sleep quality index contains 19 questions, creating 7 components that produce one global score. Higher scores indicate poorer sleep quality.
Lumbar spine range of motion | Change from Baseline (pre-treatment) to after completion of 3 months of aerobic exercise training (post-treatment)
  Lumbar spine range of motion into forward, backward, and side bending will be assessed with two inclinometers or a tape measure. subjects will

CONTACTS AND LOCATIONS:
Overall Officials: Neena Sharma, PT, PhD, CMPT, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No